CLINICAL TRIAL: NCT04821999
Title: Diode Laser 940 nm in Management of Loss of Taste Sensation in Patients With Post SARS-CoV 2 Infection
Brief Title: Diode Laser 940 nm in Management of Loss of Taste Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Alshaimaa Ahmed shabaan, associate professor in oral & maxillofacial Surgery Department, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Laser SARS-CoV2
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: SARS-CoV Infection
Keywords: SARS-CoV; , loss of taste; , Diode laser
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Ageusia | interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: Patients with SARS-CoV2 infection confirmed with PCR with loss of taste sensation
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Experimental): a 940-nm diode laser (EPIC™, BIOLASE, www.biolase.com) with an adjustable pain therapy handpiece capable of creating diffuse laser energy patterns ranging from 15 mm to 30 mm in size.
  Interventions: Device: a 940-nm diode laser
- group II (No Intervention): No treatment

INTERVENTIONS:
Device: a 940-nm diode laser — a 940-nm diode laser (EPIC™, BIOLASE, www.biolase.com) with an adjustable pain therapy handpiece capable of creating diffuse laser energy patterns ranging from 15 mm to 30 mm in size.
  Arms: group I

SUMMARY:
The global pandemic has recently emerged by transmission of SARS-CoV2 virus. The virus has had a massive impact on health, wealth and social aspects worldwide. Since the identification of this virus in Wuhan, China, millions of cases has been diagnosed worldwide with mortality rates ranging from 3% to 12 %

DETAILED DESCRIPTION:
'Long COVID' is emerging as a phenomenon where patients have long-term unresolved symptoms (8,9). These could be prolonged symptoms of SARS-CoV2 or a posteSARS-CoV2 syndrome for which dysfunction of smell and taste sensation has been proposed.

The proposal presents the diode laser 940 as possible treatment for the loss of taste sensation in patients with long SARS-CoV2. The effect of low levels of laser energy was first discovered by Dr Endre Mester in 1967.5 Since then it has been used for various applications in the field of medicine and dentistry and is broadly termed 'low level laser therapy'(LLLT) or 'biostimulation' or 'phototherapy'. It is defined as a 'non-thermal' laser light application using photons (light energy) from the visible and infrared spectrum for tissue healing and pain reduction (North American Association of Laser Therapy-NAALT). Several in vitro studies have demonstrated that the effects of laser light on wound healing are much greater than obtained with light from other sources, such as light-emitting diodes (LEDs).(10-13)

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of SARS-CoV2 with PCR. Age range from 18-60 years old Loss of taste sensation

Exclusion Criteria:

Pregnancy or contraceptive pills Lactation Any auto-immune disease that could affect the oral mucosa On any neoplastic therapy. Uncontrolled diabetes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
taste sensation survey | 6 weeks
  The participated patients will be assessed using the taste questionnaire using a category scale for rating taste intensity and a forced choice for identifying the taste quality of each sample ( salty, sweet and bitter).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halboub E, Al-Maweri SA, Alanazi RH, Qaid NM, Abdulrab S. Orofacial manifestations of COVID-19: a brief review of the published literature. Braz Oral Res. 2020 Oct 30;34:e124. doi: 10.1590/1807-3107bor-2020.vol34.0124. eCollection 2020. PMID 33146320